CLINICAL TRIAL: NCT00452166
Title: Rosiglitazone and Insulin Resistance in Renally Impaired Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: it was not possible to recruit new patients anymore
Sponsor: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p06-108a
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Last update posted 2008-10-02 (Estimated); Status verified 2008-09

CONDITIONS: Chronic Kidney Disease; Insulin Resistance
MeSH Terms: conditions — Renal Insufficiency, Chronic; Insulin Resistance | interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: rosiglitazone

SUMMARY:
30 non-diabetic, non-obese patients with stage 4 chronic kidney disease will be asked to participate in this metabolic study.

The primary aim of this study is to determine the effect of rosiglitazone on insulin resistance in non-obese patients with non-diabetic stage 4 CKD.

Secondary end points are the effects on inflammation (hsCRP), lipid profile, bone density and body composition.

DETAILED DESCRIPTION:
This part of the study will be performed in 30 non-diabetic non-obese patients. In this study patients will receive single-dose oral placebo and rosiglitazone once daily to be taken in the morning. During the first 8 weeks the patients will be dosed with 4 mg rosiglitazone. Then the concentration of the serum transaminases will be checked and if these are within an acceptable range, the doses will be doubled for the remainder of the study. If the changes in serum transaminases are considered clinically significant the patient will be withdrawn from the study and if the transaminases have increased but not to clinically significant level then the treatment of patient may be continued on the 4 mg daily dose.

The insulin sensitivity will be measured by using a euglycaemic hyperinsulinaemic clamp technique, which is validated technique.

Screening of eligible patients: fasting glucose ≤ 7,0 mmol/L and BMI ≤ 30.

Exclusion criteria are:

* A diagnosis of diabetes mellitus for which the patient uses insulin;
* Significant co-morbidities which, according to the treating nephrologists, makes it unlikely that the patient will be able to complete the foreseen study period;
* Significant cardiovascular co-morbidities which are likely to interfere with the objectives of the study (morbid obesity, family history of dyslipidemia, etc.); at the discretion of the treating nephrologists or the principal investigator;
* Allergy for PPAR's;
* Cardiac disease with marked limitation of functional capacity (New York Heart Association III or IV clinical status);
* Use of immunosuppressant agents;
* History of renal transplant;
* Hepatic insufficiency (defined as transaminase concentrations above > 2.5 times the upper limit of normal for the laboratories);
* A history of alcohol abuse or excessive alcohol use defined as more than 21 consumptions per week;
* For female patients: pregnancy, the intention to become pregnant within the study period, or lactating patients Eligible patients will receive insulin (Actrapid; Novo Nordisk A/S, Copenhagen, Denmark) at an infusion rate of 40 mU (288 pmol)/kg/m2 body surface area per minute. Euglycemia (target blood concentration of 5 mM) will be maintained by adjusting the rate of 20% glucose infusion according to whole blood glucose concentration measured from arterialized venous blood; the patient keeps his or her right arm in a box containing heated air (60°C). Insulin and glucose will be infused in the left arm. In healthy subjects, hepatic glucose production is completely suppressed when the serum insulin level is >60 mU/L. Here the expected insulin level in serum is 80 mU/L. Blood samples will be drawn at 5 min intervals for the determination of blood glucose, and at 10 min intervals during the period of 90 -120 min for the determination of serum insulin and free fatty acids. The insulin-sensitivity index (ISI) will be calculated by dividing the average glucose-infusion rate by the mean steady-state serum insulin levels during a period of 90 -120 min. In addition to glucose-infusion rate and insulin sensitivity index, the influence of the clamp on levels of FFA will also be assed.

At baseline and during the follow-up of the study inflammatory parameters (hsCRP) and lipids will be measured. At baseline and at the end a bone densitometry (DEXA) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 4
* BMI ≤ 30
* Fasting glucose < 7 mmol/l

Exclusion Criteria:

Exclusion of patients will take place in case of:

* A diagnosis of diabetes mellitus for which the patient uses insulin
* Significant co-morbidities which, according to the treating nephrologists, makes it unlikely that the patient will be able to complete the foreseen study period
* Significant cardiovascular co-morbidities which are likely to interfere with the objectives of the study (morbid obesity, family history of dyslipidemia, etc.); at the discretion of the treating nephrologists or the principal investigator
* Allergy for PPAR's
* Cardiac disease with marked limitation of functional capacity (New York Heart Association III or IV clinical status)
* Use of immunosuppressant agents
* History of renal transplant
* Hepatic insufficiency (defined as transaminase concentrations above > 2.5 times the upper limit of normal for the laboratories)
* A history of alcohol abuse or excessive alcohol use defined as more than 21 consumptions per week
* For female patients: pregnancy, the intention to become pregnant within the study period, or lactating patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-04; Primary Completion 2008-03 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 12 weeks

SECONDARY OUTCOMES:
inflammation | 12 weeks
lipid profile | 12 weeks
bone density | 12 weeks
body composition | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: andre gaasbeek, md, Principal Investigator — LUMC leiden
Locations (1):
- LUMC, Leiden, Netherlands